CLINICAL TRIAL: NCT03606031
Title: Observational Study in Patients Receiving a Digestive Microbiota Transplant According to a Standardized Protocol
Brief Title: Digestive Microbiota Transplant
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-26
Record Dates: First submitted 2018-06-27; First posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-06

CONDITIONS: Clostridium Difficile; Antibiotic Resistant Infection; Chronic Diarrhea of Unknown Origin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The digestive microbiota graft is performed in three clinical circumstances:

Clostridium difficile colitis is responsible for numerous deaths each year showing a severe prognosis. In 2013, fecal microbiote (or digestive microbiota) transplantation showed its superiority compared to the reference treatment in recurrences of C. difficile colitis. Our team has demonstrated the value of early grafting in C. difficile-associated colitis associated with ribotype 027. This strain is associated with severe cases and high mortality. In view of the major benefit observed in these particular clinical situations, investigators have implemented since 2013 in C. difficile O27 colitis and then in 2014 in severe C. difficile colitis and since May 2016 for all patients. More than 100 transplants were performed in the department dividing the risk of mortality by 5. The investigators also demonstrated the value of early fecal grafting in severe colitis irrespective of the ribotype involved. In addition, The investigators want to evaluate our protocol of fecal microbiote transplant from the first episode of C. difficile colitis in the "Unit of contagion at IHU".

2- Antibiotic-resistant bacteria In the case of digestive colonization with emergent multi-resistant bacteria, the fecal transplant has proved its effectiveness..

3- Chronic diarrhea without etiologies Finally, and after the other etiologies have been eliminated, the fecal graft may be used in this indication.

The purpose of this study is to study the characteristics of patients who have undergone treatment by grafting of digestive microbiota according to a protocol standardized either by nasogastric tube or by freeze-dried digestive microbiota capsules in 3 indications: clostridium difficile Diarrhea, multidrug resistance bacteria and chronic unexplained diarrhea without altering patient management elsewhere.

200 patients (adults) hospitalized for an episode of C. difficile colitis, multidrug resistant bacteria or chronic diarrhea without etiologies will be recruited during a period of 3 Years.

After treatment by grafting of digestive microbiota, and after signed consent, data were collected during their hospitalization and followed up at one month, 3 months, 6 month and 2 years. Data were analysed in order to determine the characteristics of patients benefiting from a digestive microbiota transplant according to a standardized protocol.

DETAILED DESCRIPTION:
The digestive microbiota graft is performed in three clinical circumstances:

1. Clostridium difficile colitis is responsible for 15,000 deaths each year in the USA. The prognosis is very severe in patients > 65 years old. In France, there were 1,800 deaths related to this infection in 2014. In 2013, fecal microbiote (or digestive microbiota) transplantation showed its superiority compared to the reference treatment in recurrences of C. difficile colitis in a randomized trial. Our team has demonstrated the value of early grafting in C. difficile-associated colitis associated with ribotype 027. This strain is associated with severe cases and high mortality. In view of the major benefit observed in these particular clinical situations, investigators have implemented since 2013 in C. difficile O27 colitis and then in 2014 in severe C. difficile colitis and since May 2016 for all patients. More than 100 transplants were performed in the department dividing the risk of mortality by 5. The investigators also demonstrated the value of early fecal grafting in severe colitis irrespective of the ribotype involved. In addition, the investigators want to evaluate our protocol of fecal microbiote transplant from the first episode of C. difficile colitis in the "Unit of contagion at the Timone IHU".
2. Antibiotic-resistant bacteria In the case of digestive colonization with emergent multi-resistant bacteria, the fecal transplant has proved its effectiveness both in the literature and in our unit.
3. Chronic diarrhea without etiologies Finally, and after the other etiologies have been eliminated, the fecal graft may be used in this indication.

The purpose of this study is to study the characteristics of patients who have undergone treatment by grafting of digestive microbiota according to a protocol standardized either by nasogastric tube or by freeze-dried digestive microbiota capsules in 3 indications: clostridium difficile Diarrhea, multidrug resistance bacteria and chronic unexplained diarrhea without altering patient management elsewhere.

200 patients (adults) hospitalized for an episode of C. difficile colitis, multidrug resistant bacteria or chronic diarrhea without etiologies will be recruited during a period of 3 Years.

After treatment by grafting of digestive microbiota, and after signed consent, data were collected during their hospitalization and followed up at one month, 3 months, 6 month and 2 years. Data were analysed in order to determine the characteristics of patients benefiting from a digestive microbiota transplant according to a standardized protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized for an episode of C. difficile colitis
* Patient hospitalized multidrug resistant bacteria
* Patient hospitalized for chronic diarrhea without etiologies
* Patient is more than 18 years old.

Exclusion Criteria:

Minor patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient hospitalized for an episode of C. difficile colitis or multidrug resistant bacteria or chronic diarrhea without etiologies
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-03-23 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
graft indications | 1 days
  * Clostridium difficile diarrhea
  * Carriage of antibiotic-resistant bacteria
  * Unexplained chronic diarrhea
recidive events | 6 months
  evolutive data will be collected in the 6 month period of follow-up
  Data will be collected during clinical consultations:
  re-hospitalization new infectection death

SECONDARY OUTCOMES:
Duration of hospitalization | up to 3 months
  beginning and end of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: EMILE GARRIDO PRADALIE, Study Director — APHM
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, PACA, France